CLINICAL TRIAL: NCT01621737
Title: Antipsychotic Effects of Oxytocin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Break in funding
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Feifel, Professor of Psychiatry and Neurosciences Program Director, Neuropsychiatry and Behavioral Medicine Program Director, UCSD Adult ADHD Program, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111017; R34MH091285 (NIH); NCT01987050 (obsolete NCT alias)
Record Dates: First submitted 2012-06-03; First posted 2012-06-18 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Schizophrenia
Keywords: oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxytocin: Low Dose (Experimental): 42 IU BID for the six weeks
  Interventions: Drug: Oxytocin
- Oxytocin: High Dose (Experimental): 84 IU BID for six weeks
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 42 IU BID for six weeks
  Arms: Oxytocin: Low Dose
Drug: Oxytocin — 84 IU BID for six weeks
  Arms: Oxytocin: High Dose
Drug: Placebo — Vehicle placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to compare the efficacy of intranasal oxytocin versus intranasal placebo to improve symptoms in schizophrenia patients who have residual symptoms despite being on adequate treatment with antipsychotic medication.

DETAILED DESCRIPTION:
This is two-site clinical study taking place at UCSD and UCI. Approximately 71 patients at each site will be randomly assigned to either intranasal oxytocin or vehicle placebo at this site.

The total duration for each individual subject will be 6 weeks on study medication (placebo or oxytocin).

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women, 21 years of age or older.
* Meet DSM-IV criteria for Schizophrenia.
* Women of childbearing potential must test negative for pregnancy at the time of enrollment based on urine pregnancy test and agree to use a reliable method of birth control during the study.
* Must be on a therapeutic dose of an atypical antipsychotic medication (examples but not limited to Clozapine Olanzapine, Risperidone, Ziprasidone, Aripiprazole, Seroquel) with no major dose changes for at least 4 weeks.
* A minimum PANSS total score of 55 at screening and baseline and a score of at least 4 (moderate) on the subscale of the PANSS (suspiciousness/persecution) at screening.
* Have a Clinical Global Impressions-Severity (CGI-S) scale score of at least 4 (moderately ill) at baseline.
* Must be able to communicate effectively with the investigator and study coordinator and have the ability to provide informed consent.
* Must be able to use nasal spray.
* Must demonstrate an acceptable degree of compliance with medication and procedures in the opinion of the investigator.

Exclusion Criteria:

* Are pregnant or are breastfeeding (negative pregnancy test at screening).
* A urine drug screen performed at screening must not show evidence of recent use of drugs of abuse.
* Any active medical condition that in the opinion of the investigator will interfere with the objectives of the study.
* Are unsuitable in any way to participate in this study, in the opinion of the investigator.
* Another current DSM-IV diagnosis other than Schizophrenia.

Permitted:

* Subjects on one SSRI, and/or sleep medication (diphenhydramine, zolpidem, zaleplon, or diazepam), at a reasonable dose, as judged by the investigator, is permitted in this study. Minor adjustments in sleep medication are acceptable. Patients will be asked to notify the study doctor of any changes to sleep aids.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Feifel, MD, Ph.D, Principal Investigator — UCSD; Steven Potkin, MD, Principal Investigator — UCI
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - University of California, San Diego, San Diego, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Groups:
- All Participants: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Period: Overall Study
Arm/Group | All Participants
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Score in the Positive and Negative Syndrome Scale (PANSS)From Baseline to Endpoint
Description: The three subscales of the PANSS include the Positive scale (7 items), the Negative scale (7 items), and the General Psychopathology scale (16 items). The total PANSS score is the sum of all 30 items of which each item is scored on a 1-7 rating system (7 indicating the worst symptoms). The items on the PANSS focus on symptoms that are common in patients with psychotic disorders and include hallucinations, delusions and disorganization as well as mood disturbances.
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: The GAF considers psychological, social, and occupational functioning on a hypothetical continuum of mental health illness. Scores on the GAF range from 1 (extremely severe) to 100 (superior functioning).
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Global Impression-Severity of Illness (CGI-S)
Description: The CGI-S is used to evaluate changes in overall severity of illness. Scores range from 1 (not at all) to 7 (among the most extremely ill).
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Clinical Global Impression-Global Improvement (CGI-I)
Description: The CGI-I is a global assessment to evaluate the subject's improvement or worsening from baseline. Scores on the CGI-I scale range from 1 (very much improved) to 7 (very much worse).
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Computerized Multiphasic Interactive Neurocognitive DualDisplayTM System (CMINDS®)
Description: The CMINDS ® consists of "construct-equivalent computerized versions of the neurocognitive assessment instruments constituting the MATRICS™ Consensus Cognitive Battery (MCCB™).
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Mayer-Salovey-Caruso Emotional Intelligence Test: Managing Emotions (MSCEIT™ ME)
Description: The MSCEIT™ ME is a multiple choice test that asses how individuals manage their emotions.
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Calgary Depression Scale for Schizophrenia (CDSS)
Description: The CDSS is a ten item diagnostic questionnaire intended to assess the severity of depression symptoms experienced by a given patient.
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Hamilton-Anxiety Scale (HAM-A)
Description: The HAM-A is a clinician administered scale for the evaluation of anxiety symptoms. It consists of 14 items of which each item is scored 0 (not present) to 4 (very severe).
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Paranoid Thoughts Scale (PTS)
Description: The PTS is a self-rated scale to assess current paranoia symptoms. The PTS consists of 32 items that the subject rates from 1 (not at all) to 5 (totally).
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: The TSMQ is a brief questionnaire asking patients about how satisfied they were with the ease, timing, etc. of the study medication giving a good indication of adherence
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Childhood Trauma Questionnaire (CTQ)
Description: The CTQ is a validated measure of adverse early experiences characterized on a measure of Anxiety Sensitivity Index and retrospective childhood maltreatment. A 5-point frequency of occurrence scale is utilized: (1) never true, (2) rarely true, (3) sometimes true, (4) often true, and (5) very often true. Each sub-scale score ranges from 5 (no history of abuse or neglect) to 25 (very extreme history of abuse and neglect).
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Experience Close Relationships (ECR)
Description: The ECR is a self-rated questionnaire designed to assess individual differences with respect to attachment-related anxiety (i.e., the extent to which people are insecure vs. secure about the extent to which their partner's availability and responsiveness) and attachment-related avoidance (i.e., the extent to which people are uncomfortable being close to others vs. secure depending on others) .
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Arizona Sexual Experience Scale (ASEX)
Description: The ASEX is a self-rated scale to assess sexual functioning. The ASEX consists of 5 items that the subject will rate from 1 ("extremely strong", "easily", or "satisfying") to 6 ("absent" or "never") based on how he/she feels at the time.
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

14. Secondary Outcome: Social Phobia Inventory (SPIN)
Description: The SPIN is a patient self-report scale that measures the degree of social phobia in a variety of different social situations.
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

15. Secondary Outcome: Penn Emotion Recognition Test (ER-40)
Description: The ER-40 is a computerized emotion discrimination test presenting 40 color photographs of evoked happy, sad, anger, fear and neutral expressions balanced for poser gender and ethnicity.
Time Frame: 6 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT01621737/Prot_SAP_000.pdf